CLINICAL TRIAL: NCT02972190
Title: Clinical Study of Bilateral Decompression With Interbody Fusion for Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Xiaofei Cheng, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNPHO-161107
Record Dates: First submitted 2016-11-07; First posted 2016-11-23 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Lumbar Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis | interventions — Laminectomy; Apoferritins; Pedicle Screws

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Bilateral decompression with TLIF (Experimental): Patients undergoing bilateral decompression with TLIF
  Interventions: Procedure: Bilateral decompression with TLIF; Device: Pedicle screw and interbody cage
- laminectomy with PLIF (Active Comparator): Patients undergoing laminectomy with PLIF
  Interventions: Procedure: laminectomy with PLIF; Device: Pedicle screw and interbody cage

INTERVENTIONS:
Procedure: Bilateral decompression with TLIF — Bilateral decompression of neural elements combined with TLIF
  Arms: Bilateral decompression with TLIF
Procedure: laminectomy with PLIF — Decompression of neural elements using laminectomy combined with PLIF
  Arms: laminectomy with PLIF
Device: Pedicle screw and interbody cage — Pedicle screw and interbody cage

SUMMARY:
Laminectomy with PLIF has been shown to achieve satisfactory clinical outcomes, but it leads to potential adverse consequences associated with extensive disruption of posterior bony and soft-tissue structures. The investigators plan to compare the clinical and radiographic outcomes of bilateral decompression with transforaminal lumbar interbody fusion and laminectomy with posterior lumbar interbody fusion in the treatment of degenerative spondylolisthesis.

ELIGIBILITY:
Inclusion Criteria:

1. lumbar spondylolisthesis
2. symptoms of low back pain and/or neurogenic claudication with or without radiculopathy referable to the lumbar spine,
3. at least 3 months of failed conservative therapies

Exclusion Criteria:

1. multilevel lumbar degenerative diseases
2. history of previous lumbar surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
visual analog scale for low back pain and leg pain | 2 years postoperatively
Oswestry disability index | 2 years postoperatively
Zurich claudication questionnaire | 2 years postoperatively
SF-36 score | 2 years postoperatively
Fusion rate | 2 years postoperatively

SECONDARY OUTCOMES:
Surgery procedure duration | Intraoperation
Estimated blood loss | Intraoperation
Length of postoperative hospital stay | 1 week after hospital discharge
Complication | 2 years postoperatively
Degree of spondylolisthesis measured by X ray | 2 years postoperatively
Disc space height measured by X ray | 2 years postoperatively
Lumbar lordosis measured by X ray | 2 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic Surgery, Shanghai Ninth People's Hospital, Shanghai, China